CLINICAL TRIAL: NCT06669832
Title: Digital Monitoring in Cancer Survivors: a Feasibility Pilot Combining a Smartwatch and Patient-reported Outcome Measures
Brief Title: Digital Monitoring in Cancer Survivors
Acronym: DM-CS
Status: Recruiting | Type: Observational
Sponsor: Laura Longshaw (Other Government)
Collaborators: Bangor University (Other); Open University (Other)
Responsible Party: Sponsor-Investigator, Laura Longshaw, Deputy Research and Development Manager, Betsi Cadwaladr University Health Board
Organization: Betsi Cadwaladr University Health Board (Other Government)
Other Study IDs: IRAS301068; IRAS 301068 (Other: Betsi Cadwaladr University Health Board)
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Digital Monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer surviviors: Cancer Survivors who are on a scheduled therapeutic break or having completed cancer treatments,

SUMMARY:
Digital monitoring in cancer survivors WHY? There is a large amount of evidence to suggest that addressing a cancer patients' quality of life and symptoms has a positive impact on their wellbeing and experience with care. Finding ways of accurately and timely measuring Patient Reported Outcomes (PROs), along with developing electronic and mobile health (eHealth and mHealth) solutions, is being increasingly recognized as one way to manage patients' quality of life and symptoms without increasing burden on time and resource-stretched National Health Services.

WHAT? The main objective of this study is to assess the feasibility of administering routine self assessment through questionnaire called the Edmonton Symptom Assessment System (ESAS) via MS Forms associated with continuous wearing of a smart watch in cancer survivors. We also hope to identify predictors of attrition or dissatisfaction.

WHO? Adult outpatients with controlled cancer undergoing surveillance (cancer survivors) WHERE? Participants will be identified through attendance in oncology outpatient clinics by the oncologist in charge.

HOW? Participants will receive a smart watch and smart phone (or an App downloaded onto their own phone). The smart watch will record physical activity , sleep patterns and other data such as heart rate and participants are expected to wear the watch all the time for about 4 months. Participants will also attend the hospital for a research appointment at the start and the end of the research and complete questionnaires weekly throughout the study, delivered via MS forms. At the end of the study the patients will be invited to a focus group to discuss their experience. The study will last for 18 months; each participants' involvement will be for about 4 month.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of any solid malignancy, at any stage

  * Completion of treatment (including surgery, radiotherapy, and any kind of cytotoxic systemic anticancer treatment [hormonal and targeted treatments allowed])
  * Clinical, biochemical and radiological confirmation of controlled disease (no evidence of residual disease or not-progressive disease)
  * Scheduled for either a therapeutic break (from cytotoxic systemic anticancer treatment), or having completed the planned multimodal treatment
  * Scheduled for active surveillance plan within oncology service or discharged to surgical or GP care following completion of adjuvant treatment
  * Male or female patients aged at least 18 years old
  * WHO Performance Status 0-2

Exclusion Criteria:

* • Not in possession of a SIM card

  * No internet access through Wi-Fi or unwilling to use mobile data allowance on a daily basis
  * Unable to understand and follow the instructions autonomously
  * Uncontrolled severe comorbidities (I.e., cardiovascular, neurological, respiratory)
  * Lack of capacity
  * Unable to understand English
  * Still undergoing systemic anticancer treatment (apart from bone-targeted agents, hormonal treatment against breast or prostate cancers or maintenance monoclonal antibody monotherapy)
  * Poor general condition (PS>2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer survivors who received treatment at Ysbyty Gwynedd, North Wales, UK.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of routine self assessment | From enrolment until end of study at 16 weeks.
  To assess the feasibility of routine self-assessment through questionnaire (ESAS) on an App associated with continuous wearing of a smart watch in cancer survivors.

CONTACTS AND LOCATIONS:
Locations (1):
- Betsi Cadwaladr University Health board, Bangor, Gwynedd, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided